CLINICAL TRIAL: NCT06362525
Title: Incidence of Episodes of (Dis)Connected Consciousness Among Emergency Patients Admitted in the Resuscitation Room
Status: Recruiting | Type: Observational
Sponsor: University of Liege (Other)
Collaborators: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-389
Record Dates: First submitted 2023-08-29; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-06

CONDITIONS: Critical Illness; Near-Death Experience; Consciousness, Loss of; Quality of Life; Emergencies
Keywords: Dream
MeSH Terms: conditions — Critical Illness; Death; Unconsciousness; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to describe the incidence of episodes of disconnected consciousness (including near-death experience (NDE)) and episodes of connected consciousness in patients admitted to the resuscitation room, who survived a critical condition and who meet at least one of these criteria during their stay in the resuscitation room: (1) deep sedation, (2) intubation, (3) cardiopulmonary resuscitation, or (4) (non-drug-induced) Glasgow Coma Scale score = 3. We also investigate the potential (neuro)physiological markers and biomarkers. In order to help determine the potential risk factors of such episodes, cognitive factors such as dissociative propensity are also investigated. Unexpected visual and auditory stimuli will be displayed. In addition, we assess the evolution of memory, as well as short- and long-term consequences on quality of life, anxiety, and attitudes towards care.

Memory of patients who did not meet the above-mentioned criteria are also investigated. A group of 15 healthy participants will be invited to test the stimuli display.

Finally, (neuro)physiological parameters of a subsample of dying patients are also investigated.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted in the resuscitation room of our university hospital
* French speaking

Exclusion Criteria:

* Refusal
* Chronic disorder of consciousness
* Deafness
* Blindness
* Dementia
* Hemineglect
* Aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted in the resuscitation room
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Detection of potential episodes of disconnected consciousness | upon awakening/discharge from the resuscitation room (max 21 days after the admission in the room)
  near-death experience (using the Near-Death Experience Content scale); dream
Detection of potential episodes of connected consciousness | upon awakening/discharge from the resuscitation room (max 21 days after the admission in the room)
  explicit recall of environmental/external stimuli upon awakening

SECONDARY OUTCOMES:
Risk factors | in the resusctiation room admission
  (neuro)physiological marker; biomarker; cognitive factor
Quality of life assessment | at 6-month
  The EuroQol five-dimension three-level questionnaire (EQ-5D-3L) comprises two sections. The first one is a five-question descriptive component which explores five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each question has three possible answers, rated from 1 to 3 (no problems, some problems and extreme problems). The second section is a visual analogue scale (EQ VAS; 0 "worst imaginable health state" to 100 "best imaginable health state") about their current health state.
Memory content and evolution assessment | at 1-month
  The Memory Characteristics Questionnaire (MCQ). A total score can be derived summing all the 16 items (each on a 1-7 points Likert scale) and refers to as the amount of memory characteristics (i.e. higher total scores reflect greater amount of memory characteristics).
Detection of post-traumatic stress disorder (PTSD) | at 6-month
  The Posttraumatic Stress Disorder Checklist 5 (PCL-5). Its total score can range from 0 to 80 (scores of ≥31 suggest a probable diagnosis of PTSD)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data will be anonymized and shared among collaborators upon reasonable request and agreement
Supporting Information: Study Protocol
Time Frame: Data will be shared with collaborators for the specified time allocated to each respective project. Whereas, data shared on the database will be anonymized and available indefinitely.
Access Criteria: A written agreement between the groups (university or research teams)